CLINICAL TRIAL: NCT03431415
Title: Surgery Versus Stereotactic Body Radiation Therapy for Stage up to IA2 (T1a or T1b) Non-small Cell Lung Cancer
Acronym: RAXSIA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual issues
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Paula Antonia Ugalde Figueroa, Research Coordinator (Thoracic Surgery), Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAXSIA
Record Dates: First submitted 2018-01-28; First posted 2018-02-13 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Non-small Cell Lung Cancer Stage I; Surgery; Stereotactic Body Radiation Therapy
Keywords: Lung; Cancer; Early-Stage; Video-assisted Thoracic Surgery; VATS; SBRT; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Active Comparator): Patients that will undergo surgery (anatomical segmentectomy, lobectomy or bilobectomy) as primary lung cancer treatment
  Interventions: Procedure: Anatomical Segmentectomy, Lobectomy or Bilobectomy
- SBRT (Stereotactic Body Radiation Therapy) (Active Comparator): Patients that will undergo SBRT as primary lung cancer treatment
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Anatomical Segmentectomy, Lobectomy or Bilobectomy — Lung Cancer Anatomical Resection
  Arms: Surgery
Radiation: Stereotactic Body Radiation Therapy — SBRT treatment. 48Gy in 4 sessions for peripheral lesions and 50Gy in 5 sessions for central lesions.
  Arms: SBRT (Stereotactic Body Radiation Therapy)

SUMMARY:
The primary objective of this study is disease free survival rate at 5 years in stage IA2 (T1aN0M0 or T1bN0M0 only) non-small cell lung cancer (NSCLC) patients treated either by surgery or stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
Today, the best medical literature available confirms that surgery is superior to radiation therapy in the treatment of the early stage lung cancer. However, good emerging data demonstrates potential equality between these two treatments. Two major international studies have tried to compare both treatments but have failed to complete the study because of the lack of patients accrual. We chose to design a trial in which patients will be part of a shared decision making process in selecting the treatment modality.

Patients with early stage lung cancer, that can undergo surgical treatment will be offered SBRT, and in conjunction with the pulmonologist will decide which treatment they prefer. We intend to complete the recruitment of patients within 02 years, then follow-up for 5 more years to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75
* Pathologically (histologically or cytologically) proven NSCLC.
* Stage IA2 T1aN0M0 or T1bN0M0 only, fit for surgery.

  * Tumor ≤ 2 cm (T1a or T1b according to AJCC, 8th ed.)
* Hilar or mediastinal lymph nodes ≤ 1 cm with no abnormal hilar or mediastinal uptake on PET scan are considered N0.

  * Patients with hilar or mediastinal lymph nodes > 1 cm on CT scan or abnormal PET scan (including suspicious but non-diagnostic uptake) are eligible, provided directed tissue biopsies by EBUS or mediastinoscopy of all abnormally identified areas are negative for cancer.
  * EBUS preferable
  * No regional or distant metastases.
* Resectable disease and treatable by SBRT
* Peripherally located tumor.

  * Primary tumor within or touching the zone of the proximal bronchial tree, defined as a volume of 2 cm in all directions around the proximal bronchial tree are excluded (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi).
  * No involvement of the central pleura and/or structures of the mediastinum.
* Staging studies must be done within 8 weeks prior to study entry
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Previously operated lung cancer.
* Previous thoracic irradiation.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
* Pulmonary nodule manifested as pure ground-glass opacity.
* Severe pulmonary hypertension.
* Severe cardiac, hepatic or renal insufficiency.
* Severe peripheral vascular disease.
* Severe cerebral or psychiatric pathologies.
* Severe chronic heart disease.
* Life expectancy < 6 months.
* Pregnant or lactating woman.
* Unwilling to have follow-up.
* Central tumor where pneumonectomy might be considered.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  To compare the disease free survival of patients with Stage up to IA2 (T1aN0M0 or T1bN0M0) NSCLC managed either by SBRT or surgery.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall survival rate at 5 years in both arms
Level of morbidity | 5 years
  Level of morbidity in both arms (CTCAE 4.0 - common toxicity criteria)
Level of efficacy in the SBRT arm | 5 years
  Level of efficacy in the SBRT arm (RECIST 1.1)
QOL assessment | 5 years
  QOL assessment with SF36 questionnaire (pre and post treatment) in both arms
FEV1 and DLCO decline at 1-year post-treatment in both arms | 1 year
  FEV1 or DLCO decline at 1-year post-treatment in both arms
Health economic evaluation in both arms | 5 years
  Health economic evaluation in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Ugalde Figueroa, MD, Principal Investigator — Associate Professor, Thoracic Surgeon, Research Coordinator
Locations (2):
- Canada (2):
  - Hôtel-Dieu de Québec (CHUQ), Québec, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec - Université Laval, Québec, Quebec